CLINICAL TRIAL: NCT02379481
Title: Effects of Deer Bone Extract NS on Improvement in Cognitive-Bio-Markers of Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT_NS
Record Dates: First submitted 2014-03-27; First posted 2015-03-05 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Adults With Subjective Memory Complaints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- NS 550mg (Experimental): NS 550mg/day
  Interventions: Dietary Supplement: NS 550mg
- NS 1100mg (Experimental): NS 1100mg/day
  Interventions: Dietary Supplement: NS 1100mg
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: NS 550mg
  Arms: NS 550mg
Dietary Supplement: NS 1100mg
  Arms: NS 1100mg
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
This study aims to elucidate the effects of deer bone extract NS on cognitive function improvement and its safety in healthy adults aged 40 to 65 years who report decline in subjective cognitive functions using multimodal neuroimaging and neurocognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years old,
* Global Deterioration Scale score (GDS) of 2
* High school or higher levels of education.

Exclusion Criteria:

* Current pregnancy or breast-feeding
* Evidence of neurologic or medical conditions
* Axis I diagnosis when assessed by the board certified psychiatrist using the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorder, 4th edition (DSM-IV)(SCID-IV),
* One or more major depressive episode during last 12 months
* Mini-mental status examination score of 24 or less
* Clinical Dementia Rating score of 0.5 or more suggesting cognitive impairment beyond self-perceived subjective deficits
* Intelligence quotient less than 70
* Any history of head trauma involving loss of consciousness or seizure
* Contraindications to magnetic resonance imaging (MRI)
* Use of psychotropics in last 3 months
* Use of oral contraceptive medication
* Participation in other clinical trials during the study period that might affect the outcome of the present study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in neurocognitive function | Baseline, 8th week
  Scores from neurocognitive test batteries such as CANTAB
Changes from baseline in brain structure analyzed using the computational approach | Baseline, 8th week
  Morphometric analysis of brain structures in magnetic resonance imaging
Changes from baseline in brain function analyzed using the computational approach | Baseline, 8th week
  Blood oxygenation level dependent (BOLD) signal intensity and their connectivity assessed using functional magnetic resonance imaging scans
Changes from baseline in brain biochemical metabolism analyzed using the computational approach | Baseline, 8th week
  Brain metabolite concentrations assessed using magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Change from baseline in Subjective Memory Complaints Questionnaire scores at 8th weeks | Baseline, 8th week
Number of participants with adverse events | 1st week
Number of participants with adverse events | 4th week
Number of participants with adverse events | 8th week

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University, Seoul, South Korea

REFERENCES:
- [Derived] Jeon Y, Kim B, Kim JE, Kim BR, Ban S, Jeong JH, Kwon O, Rhie SJ, Ahn CW, Kim JH, Jung SU, Park SH, Lyoo IK, Yoon S. Effects of Ganglioside on Working Memory and the Default Mode Network in Individuals with Subjective Cognitive Impairment: A Randomized Controlled Trial. Am J Chin Med. 2016;44(3):489-514. doi: 10.1142/S0192415X16500270. Epub 2016 Apr 24. PMID 27109158